CLINICAL TRIAL: NCT01275469
Title: A Pilot Study to Evaluate the Efficacy and Safety of GFT505 (80 mg) Orally Administered Once Daily for 35 Days in Patients Presenting With Impaired Glucose Tolerance and Abdominal Obesity. A Double Blind, Parallel Group, Placebo-controlled and Randomized Study.
Brief Title: Pilot Study With GFT505 (80mg) in Patients Presenting With Impaired Glucose Tolerance and Abdominal Obesity.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genfit (Industry)
Responsible Party: Product Development Department, GENFIT
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GFT505-209-4; 2009-011003-23 (EudraCT Number)
Record Dates: First submitted 2011-01-10; First posted 2011-01-12 (Estimated); Last update posted 2011-01-12 (Estimated); Status verified 2011-01

CONDITIONS: Impaired Glucose Tolerance; Abdominal Obesity
Keywords: Impaired Glucose tolerance; OGTT; PPARs
MeSH Terms: conditions — Glucose Intolerance; Obesity, Abdominal | interventions — 2-(2,6-dimethyl-4-(3-(4-(methylthio)phenyl)-3-oxo-1-propenyl)phenoxyl)-2-methylpropanoic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- GFT505 80mg (Experimental)
  Interventions: Drug: GFT505 80mg
- Matching placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GFT505 80mg — Hard gelatin capsules dosed at 20mg, oral administration, 4 capsules per day before breakfast.
  Arms: GFT505 80mg
Drug: Placebo — Hard gelatin capsules, oral administration, 4 capsules per day before breakfast.
  Arms: Matching placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy of GFT505 80mg compared with placebo in improving Oral Glucose Tolerance Test (OGTT), in patients with impaired glucose tolerance and abdominal obesity, and to assess the tolerability and safety of once-a-day administrations of oral doses of GFT505 during 35 days.

DETAILED DESCRIPTION:
The study period is 13 weeks maximum per patient : A screening period (1 to 6-weeks) will precede a 5-week double-blind treatment period and a 2-week follow-up period. The duration of the screening period will depend on the necessity to introduce a wash-out for lipid-lowering drugs : 4-week wash-out from statins and other lipid regulating drugs and 6-week wash-out from fibrates. During the screening period, patients will be asked to start or continue adequate diet and exercise.

ELIGIBILITY:
Inclusion Criteria:

* Male or post-menopausal female.
* Waist circumference ≥94cm for male, ≥ 80cm for female.
* Fasting Plasma Glucose (FPG) between 110 and 126 mg/dl (between 6.1 and 7.0 mmol/l) within 6 months prior to the screening visit.
* 2-hour glycaemia at OGTT (2hr after a 75g oral glucose load) ≥140 mg/dL (7.8 mmol/l).

Exclusion Criteria:

* Body Mass Index (BMI) ≥ 40 kg/m².
* Blood Pressure > 160 / 95 mmHg.
* Known Type I or type II Diabetes Mellitus.
* Glycated haemoglobin (HbA1c) >7%.
* A fasting TG > 400mg/dl and a LDL-C > 220mg/dl.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2009-06; Primary Completion 2009-12 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Oral Glucose test Tolerance (OGTT) | 4 weeks
  To evaluate the change in plasma Glucose 2hr following oral glucose load from baseline to end point. Evaluation will be made during the selection period, prior any drug intake, and 4 weeks (28-34 days) after the first treatment intake.

SECONDARY OUTCOMES:
Volume oxygen maximal (VO2max) | 5 weeks
  To evaluate the efficacy of GFT505 80mg compared with placebo in improving the VO2max at physical exercise test. Evaluation will be made during the selection period, prior any drug intake, and 5 weeks after the first treatment intake.
Respiratory parameters measured during the physical exercise test | 5 weeks
  To describe the changes on others parameters measured during the physical exercise test : Volume carbon dioxide (VCO2), Respiratory quotient (RQ), Lactate concentration. Evaluation will be made during the selection period, prior any drug intake, and 5 weeks after the first treatment intake.
Fasting Glycemia and Insulinemia | 5 weeks
  To describe the changes of fasting glycaemia and insulinemia in the two groups. Evaluation will be made the first day prior any drug intake, then 5 weeks after the first treatment intake.
HOMA index (Homeostasis Model Assessment) | 5 weeks
  To describe the changes of HOMA index in the two groups. Evaluation will be made the first day prior any drug intake, then 5 weeks after the first treatment intake.
Lipids | 5 weeks
  To describe the changes in Triglycerides (TG), High Density Lipoprotein Cholesterol (HDL-C), Low Density Lipoprotein Cholesterol (LDL-C) and non High Density Lipoprotein Cholesterol (non-HDL-C) levels in the two groups. Evaluation will be made the first day prior any drug intake, then 2-3, and 4 weeks after the first treatment intake and 2 weeks after the last treatment intake (follow-up visit).

CONTACTS AND LOCATIONS:
Overall Officials: Rémy Hanf, Development Director, Study Director — GENFIT, France; Eric BRUCKERT, Pr., Study Chair — University Hospital of Paris 6, France
Locations (20):
- France (20):
  - Site n°31, Angers
  - Site n°32, Angers
  - Site n°36, Angers
  - Site n°37, Angers
  - Site n°34, Angers
  - Site n°35, Angers
  - Site n°39, Angers
  - Site n°17, Briollay
  - Site n°16, Cholet
  - Site n°19, Cholet
  - Site n°14, Le Mesnil-en-Vallée
  - Site n°10, Mûrs-Erigné
  - Site n°12, Mûrs-Erigné
  - Site n°2, Nantes
  - Site n°13, Parçay-les-Pins
  - Site n°1, Paris
  - Site n°15, Segré
  - Site n°11, Thouars
  - Site n°30, Tiercé
  - Site n°18, Vihiers

REFERENCES:
- [Derived] Staels B, Rubenstrunk A, Noel B, Rigou G, Delataille P, Millatt LJ, Baron M, Lucas A, Tailleux A, Hum DW, Ratziu V, Cariou B, Hanf R. Hepatoprotective effects of the dual peroxisome proliferator-activated receptor alpha/delta agonist, GFT505, in rodent models of nonalcoholic fatty liver disease/nonalcoholic steatohepatitis. Hepatology. 2013 Dec;58(6):1941-52. doi: 10.1002/hep.26461. Epub 2013 Oct 29. PMID 23703580
- [Derived] Cariou B, Zair Y, Staels B, Bruckert E. Effects of the new dual PPAR alpha/delta agonist GFT505 on lipid and glucose homeostasis in abdominally obese patients with combined dyslipidemia or impaired glucose metabolism. Diabetes Care. 2011 Sep;34(9):2008-14. doi: 10.2337/dc11-0093. Epub 2011 Aug 4. PMID 21816979